CLINICAL TRIAL: NCT03572075
Title: Evaluation of the Efficacy of Pelvic Floor Physiotherapy in Symptomatic Patients Affected by Deep Infiltrating Endometriosis
Brief Title: Physiotherapy of the Pelvic Floor in Women With Deep Infiltrating Endometriosis
Acronym: endofisio-01
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Mohamed Mabrouk, Principal investigator, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 345/2017/O/Sper
Record Dates: First submitted 2018-05-27; First posted 2018-06-28 (Actual); Last update posted 2019-06-12 (Actual); Status verified 2019-06

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): assessment of symptoms at the first medical examination; standard care protocol; pelvic floor physiotherapy; assessment of symptoms after four months
  Interventions: Diagnostic Test: assessment of symptoms at the first medical examination; Procedure: pelvic floor physiotherapy; Procedure: standard care protocol; Diagnostic Test: assessment of symptoms after four months
- Group B (Experimental): assessment of symptoms at the first medical examination; standard care protocol; assessment of symptoms after four months
  Interventions: Diagnostic Test: assessment of symptoms at the first medical examination; Procedure: standard care protocol; Diagnostic Test: assessment of symptoms after four months

INTERVENTIONS:
Diagnostic Test: assessment of symptoms at the first medical examination — assessment of endometriosis related symptoms using NRS (Numerical Rating Scale); intestinal, sexual and urinary functions are evaluated with validated questionnaires (Knowles-Eccersley-Scott-Symptom Questionnaire (KESS), Female Sexual Function Index (FSFI), Bristol Female Lower Urinary Tract Symptoms (BFLUTS)); pelvic floor morphometry at rest, during pelvic floor contraction and during Valsalva manoeuvre is evaluated using 3D/4D transperineal ultrasound through the assessment of the levator hiatus area (LHA) at the first medical examination
Procedure: pelvic floor physiotherapy — six individual sessions (weeks 1, 3 , 5, 8, 11 from the randomization) with pelvic floor consciousness exercises with mild contractions and relaxation (ex. 'kegel reverse' exercises); respiratory rate control exercises; extra exercises to perform at home are suggested.
  Arms: Group A
Procedure: standard care protocol — the treatment is the same as usual in our center
Diagnostic Test: assessment of symptoms after four months — assessment of endometriosis related symptoms using NRS (Numerical Rating Scale); intestinal, sexual and urinary functions are evaluated with validated questionnaires (Knowles-Eccersley-Scott-Symptom Questionnaire (KESS), Female Sexual Function Index (FSFI), Bristol Female Lower Urinary Tract Symptoms (BFLUTS)); pelvic floor morphometry at rest, during pelvic floor contraction and during Valsalva manoeuvre is evaluated using 3D/4D transperineal ultrasound through the assessment of the levator hiatus area (LHA) after four months from the randomization.

SUMMARY:
The aim of our study is to evaluate the impact of pelvic floor physiotherapy in symptomatic patients affected by deep infiltrating endometriosis, using 3D/4D transperineal ultrasound for evaluation of pelvic floor morphometry, NRS (Numerical Rating Scale) for evaluation of symptoms and validated questionnaires investigating intestinal, sexual and urinary functions.

These results will be compared with those obtained from symptomatic patients affected by deep infiltrating endometriosis following the standard care procedure that does not provide pelvic floor physiotherapy.

DETAILED DESCRIPTION:
Symptomatic, nulliparous women with deep infiltrating endometriosis are included in the study.

During the first medical examination, endometriosis related symptoms are assessed using NRS (Numerical Rating Scale); intestinal, sexual and urinary functions are evaluated with validated questionnaires (Knowles-Eccersley-Scott-Symptom Questionnaire (KESS), Female Sexual Function Index (FSFI), Bristol Female Lower Urinary Tract Symptoms (BFLUTS)); pelvic floor morphometry at rest, during pelvic floor contraction and during Valsalva manoeuvre is evaluated using 3D/4D transperineal ultrasound through the assessment of the levator hiatus area (LHA). Gynaecological examination, transvaginal and transabdominal ultrasound are performed.

After the first medical examination, enrolled patients are randomized into two groups: patients in Group A receive standard care procedure and pelvic floor physiotherapy; patients in Group B receive standard care procedure only. Pelvic floor physiotherapy protocol consists of six sessions (weeks 1, 3, 5, 8, 11 from the randomization). After four months from the first medical examination, endometriosis related symptoms, intestinal, sexual and urinary functions and pelvic floor morphometry are reassessed for all patients, using the same procedures, comparing the two groups and evaluating the impact of pelvic floor physiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical and ultrasound diagnosis of deep endometriosis with related symptoms (chronic pelvic pain, dysmenorrhea, dyschezia, dyspareunia, dysuria)
* Nulliparity
* Obtaining Informed Consent

Exclusion Criteria:

* Patients with an oncological disease or needing surgery for malignant pathologies
* Urogenital prolapse
* History of surgery for deep infiltrating endometriosis
* Congenital or acquired malformations of pelvis and pelvic floor
* History of diseases characterised by chronic pelvic pain (interstitial cystitis, irritable bowel disease, chronic vulvodynia).

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-06-15 (Actual); Primary Completion 2019-09 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the impact of pelvic floor physiotherapy on intestinal function | After four months from the randomization
  Evaluation of the impact of pelvic floor physiotherapy on symptomatic patients, using a validated questionnaire (Knowles-Eccersley-Scott-Symptom Questionnaire (KESS).
Evaluation of the impact of pelvic floor physiotherapy on sexual function | After four months from the randomization
  Evaluation of the impact of pelvic floor physiotherapy on symptomatic patients, using a validated questionnaire (Female Sexual Function Index (FSFI)).
Evaluation of the impact of pelvic floor physiotherapy on urinary function | After four months from the randomization
  Evaluation of the impact of pelvic floor physiotherapy on symptomatic patients, using a validated questionnaire (Bristol Female Lower Urinary Tract Symptoms (BFLUTS)).
Evaluation of the impact of pelvic floor physiotherapy on pelvic floor muscles contraction | After four months from the randomization
  Evaluation of the impact of pelvic floor physiotherapy on pelvic floor muscles contraction and pain using a gynecological examination and ultrasounds. All scans are obtained using a Voluson E6 system (GE Healthcare, Zipf, Austria) with RAB 8-4-MHz volume transducer for all acquisitions. Measurements were evaluated using a dedicated software (4DView 14.4; GE Healthcare, Zipf, Austria).

SECONDARY OUTCOMES:
Evaluation of uro-genital hiatus using 3D-4D transperineal ultrasound | At randomization and after four months from the randomization
  Women are firstly asked to rest and then contract the pelvic floor muscles (PFM) until the maximal cranioanterior displacement of the anorectal angle is attained.
  The anorectal angle is defined as the angle between the posterior wall of the rectal ampulla and the anal canal.
  All scans are obtained using a Voluson E6 system (GE Healthcare, Zipf, Austria) with RAB 8-4-MHz volume transducer for all acquisitions. Measurements were evaluated using a dedicated software (4DView 14.4; GE Healthcare, Zipf, Austria).
Evaluation of the 3D-4D transperineal ultrasound as a bio-feedback tool | After 1, 3, 5, 8, 11 weeks from the randomization
  Patients are firstly asked to rest and then contract the pelvic floor muscles looking at the ultrasound screen in order to be aware of the contraction of the pelvic floor muscles and improve it. Voluson E6 system (GE Healthcare, Zipf, Austria) with RAB 8-4-MHz volume transducer is used for all acquisitions.

CONTACTS AND LOCATIONS:
Locations (1):
- Gynecology and Physiopathology of Human Reproductive Unit, University of Bologna, S. Orsola-Malpighi Hospital, Bologna, BO, Italy